CLINICAL TRIAL: NCT02352714
Title: Study of Pain Control With Hormonal IUS Insertion (SOPHI Study)
Brief Title: Study of Pain Control With Hormonal IUS Insertion
Acronym: SOPHI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Bayer (Industry); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 14-011286
Record Dates: First submitted 2015-01-22; First posted 2015-02-02 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Pain
Keywords: Adolescents; Women's Health; Contraception; Reproduction; Comparative Effectiveness Research; Pregnancy Prevention; Intrauterine Device
MeSH Terms: conditions — Pain | interventions — Anesthesia, Obstetrical; Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paracervical Nerve Block (Active Comparator): Ten milliliters of 1% lidocaine paracervical anesthetic will be injected at three cervical locations: 1 mL at the tenaculum site (12 o'clock on a clock face) and 4.5 mL each at the 4 o'clock and 8 o'clock positions. A 3 minute waiting period will be used between the administration of the paracervical nerve block and the insertion of IUS to allow the paracervical block to take effect.
  Interventions: Drug: Paracervical Nerve Block
- Sham Paracervical Block (Sham Comparator): To perform the sham cervical block, the cervix will be touched with the blunt end of a Q-tip at the three locations described above for the paracervical block. The cervical mucosa will not be broken during the sham block. A 3 minute waiting period will again occur between administration of the sham block and IUS insertion to be consistent with the procedure used for the nerve block.
  Interventions: Drug: Sham Paracervical Block

INTERVENTIONS:
Drug: Paracervical Nerve Block — Block randomization to receive lidocaine paracervical nerve block vs sham cervical block
  Other Names: 1 % Lidocaine
  Arms: Paracervical Nerve Block
Drug: Sham Paracervical Block — Block randomization to receive lidocaine paracervical nerve block vs sham cervical block
  Other Names: Blunt End of a Q-Tip
  Arms: Sham Paracervical Block

SUMMARY:
This study aims to compare pain during insertion of the Skyla® IUS using a 100mm visual analog scale (VAS) among 92 young women aged 14 to 22 years randomized to receive a paracervical (n=46) block versus a sham paracervical block (n=46).

DETAILED DESCRIPTION:
Intrauterine systems (IUS) are among the most effective forms of reversible contraception. Numerous studies demonstrate their safety and efficacy. Despite this, uptake of IUSs among U.S. young women aged 14 to 22 years has been low. Increasing the use of this effective, long acting contraception among young women is an important public health goal, as it could help to reduce the high rates of unintended pregnancies in this population.

A major barrier to young women's utilization of IUSs is fear of pain during insertion. Unfortunately, studies evaluating methods of pain control during IUS insertion have focused on adult women, leaving the question unanswered as to the best pain management method for young women. Compared to adult women, young women have less experience with pelvic exams and may therefore derive greater benefit from pain control measures during gynecologic procedures, such as IUS insertions. Young women and their providers are seeking effective pain control options; yet, there is a lack of high quality, comparative effectiveness research to guide decision making. This proposal seeks to fill this important gap.

With the introduction of the Skyla IUS (Bayer Healthcare Pharmaceuticals, Inc.) to the U.S. market in January 2013, a new approach to pain management became possible. Skyla is smaller than existing IUSs and may therefore cause less pain during insertion. The pain response triggered during Skyla insertion may be better controlled by existing pain control options. This is the underlying premise of this study.

In addition to the size of an IUS, theoretical and empirical data suggest that paracervical blocks have the greatest promise for pain control during IUS insertion compared to other pain control options. Paracervical infiltration of a local anesthetic into the cervix interrupts the visceral sensory fibers of the lower uterus, cervix, and upper vagina. Data from several clinical trials indicate that paracervical blocks provide clinically significant control of pain during multiple types of gynecologic procedures. One recently published study evaluated the effectiveness of paracervical blocks during IUS insertion and found a marginally significant reduction in pain, but the study was underpowered and focused on adult women. The value of a paracervical block in young women receiving an IUS remains unclear.

The investigator propose to conduct a randomized, controlled single-blind trial comparing pain with Skyla IUS insertion among young women aged 14 to 22 years randomized to receive a paracervical block versus a sham cervical block. This study will provide important information for counseling young women about pain management during IUS insertion.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous (i.e., no pregnancy > 24 weeks)
* Not currently pregnant
* Not pregnant in the past 6 weeks
* Willing to be randomized to a paracervical nerve block or sham paracervical block group
* Interested in using an intrauterine system (IUS)
* Able to read and provide written informed consent in English

Exclusion Criteria:

* An allergy, hypersensitivity, or absolute medical contra-indication to using lidocaine, other amino-amide local anesthetics, or to non-steroidal anti-inflammatory agents, such as ibuprofen
* A history of epilepsy or peptic ulcer disease
* Moderate to severe asthma that precludes non-steroidal anti-inflammatory drug (NSAID) use
* Hepatic or renal failure
* Moderate to severe cardiac disease
* Previous use of an IUS or a history of a prior failed IUS insertion
* Use of a narcotic or benzodiazepine in the past 24 hours
* Positive pregnancy test or reasonable risk of pregnancy
* Current cervicitis
* Intrauterine infection in the past 90 days
* Meet Centers for Disease Control Medical Eligibility Criteria (MEC) category 3 or 4 classification for IUS use
* Currently breastfeeding

Ages: 14 Years to 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 98 (Actual)
Dates: Start 2015-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Self-reported pain | Intraoperative (At the time of insertion of the IUS)
  The primary outcome will be assessed using a visual analogue scale (VAS). Assessment will occur at the time of the insertion of the IUS device. The IUS will be placed according to manufacturer's recommendation.

CONTACTS AND LOCATIONS:
Overall Officials: Aletha Y Akers, MD, MPH, Principal Investigator — Children's Hospital of Philadelphia
Locations (3):
- United States (3):
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - The Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospitals, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kavanaugh ML, Jerman J, Hubacher D, Kost K, Finer LB. Characteristics of women in the United States who use long-acting reversible contraceptive methods. Obstet Gynecol. 2011 Jun;117(6):1349-1357. doi: 10.1097/AOG.0b013e31821c47c9. PMID 21606745
- [Background] Finer LB, Jerman J, Kavanaugh ML. Changes in use of long-acting contraceptive methods in the United States, 2007-2009. Fertil Steril. 2012 Oct;98(4):893-7. doi: 10.1016/j.fertnstert.2012.06.027. Epub 2012 Jul 13. PMID 22795639
- [Background] Finer LB. Unintended pregnancy among U.S. adolescents: accounting for sexual activity. J Adolesc Health. 2010 Sep;47(3):312-4. doi: 10.1016/j.jadohealth.2010.02.002. Epub 2010 Apr 9. PMID 20708573
- [Background] Kavanaugh ML, Frohwirth L, Jerman J, Popkin R, Ethier K. Long-acting reversible contraception for adolescents and young adults: patient and provider perspectives. J Pediatr Adolesc Gynecol. 2013 Apr;26(2):86-95. doi: 10.1016/j.jpag.2012.10.006. Epub 2012 Dec 31. PMID 23287602
- [Background] Hubacher D, Reyes V, Lillo S, Zepeda A, Chen PL, Croxatto H. Pain from copper intrauterine device insertion: randomized trial of prophylactic ibuprofen. Am J Obstet Gynecol. 2006 Nov;195(5):1272-7. doi: 10.1016/j.ajog.2006.08.022. PMID 17074548
- [Background] Massey SE, Varady JC, Henzl MR. Pain relief with naproxen following insertion of an intrauterine device. J Reprod Med. 1974 Dec;13(6):226-31. No abstract available. PMID 4612152
- [Background] Heikinheimo O, Inki P, Kunz M, Parmhed S, Anttila AM, Olsson SE, Hurskainen R, Gemzell-Danielsson K. Double-blind, randomized, placebo-controlled study on the effect of misoprostol on ease of consecutive insertion of the levonorgestrel-releasing intrauterine system. Contraception. 2010 Jun;81(6):481-6. doi: 10.1016/j.contraception.2010.01.020. Epub 2010 Mar 1. PMID 20472114
- [Background] Dijkhuizen K, Dekkers OM, Holleboom CA, de Groot CJ, Hellebrekers BW, van Roosmalen GJ, Janssen CA, Helmerhorst FM. Vaginal misoprostol prior to insertion of an intrauterine device: an RCT. Hum Reprod. 2011 Feb;26(2):323-9. doi: 10.1093/humrep/deq348. Epub 2010 Dec 15. PMID 21159683
- [Background] Edelman AB, Schaefer E, Olson A, Van Houten L, Bednarek P, Leclair C, Jensen JT. Effects of prophylactic misoprostol administration prior to intrauterine device insertion in nulliparous women. Contraception. 2011 Sep;84(3):234-9. doi: 10.1016/j.contraception.2011.01.016. Epub 2011 Mar 3. PMID 21843686
- [Background] Mody SK, Kiley J, Rademaker A, Gawron L, Stika C, Hammond C. Pain control for intrauterine device insertion: a randomized trial of 1% lidocaine paracervical block. Contraception. 2012 Dec;86(6):704-9. doi: 10.1016/j.contraception.2012.06.004. Epub 2012 Jul 6. PMID 22770792
- [Background] Bednarek PH, Micks EA, Edelman AB, Li H, Jensen JT. The effect of nitroprusside on IUD insertion experience in nulliparous women: a pilot study. Contraception. 2013 Apr;87(4):421-5. doi: 10.1016/j.contraception.2012.10.030. Epub 2012 Dec 4. PMID 23218853
- [Background] McNicholas CP, Madden T, Zhao Q, Secura G, Allsworth JE, Peipert JF. Cervical lidocaine for IUD insertional pain: a randomized controlled trial. Am J Obstet Gynecol. 2012 Nov;207(5):384.e1-6. doi: 10.1016/j.ajog.2012.09.018. Epub 2012 Sep 20. PMID 23107081
- [Background] Tangsiriwatthana T, Sangkomkamhang US, Lumbiganon P, Laopaiboon M. Paracervical local anaesthesia for cervical dilatation and uterine intervention. Cochrane Database Syst Rev. 2009 Jan 21;(1):CD005056. doi: 10.1002/14651858.CD005056.pub2. PMID 19160245
- [Background] Ahmad G, Duffy J, Watson AJ. Pain relief in hysterosalpingography. Cochrane Database Syst Rev. 2007 Apr 18;(2):CD006106. doi: 10.1002/14651858.CD006106.pub2. PMID 17443612
- [Background] Renner RM, Jensen JT, Nichols MD, Edelman AB. Pain control in first-trimester surgical abortion: a systematic review of randomized controlled trials. Contraception. 2010 May;81(5):372-88. doi: 10.1016/j.contraception.2009.12.008. Epub 2010 Jan 27. PMID 20399943
- [Background] Karabayirli S, Ayrim AA, Muslu B. Comparison of the analgesic effects of oral tramadol and naproxen sodium on pain relief during IUD insertion. J Minim Invasive Gynecol. 2012 Sep-Oct;19(5):581-4. doi: 10.1016/j.jmig.2012.04.004. Epub 2012 Jul 4. PMID 22766124
- [Background] Jensen HH, Blaabjerg J, Lyndrup J. [Prophylactic use of prostaglandin synthesis inhibitors in connection with IUD insertion]. Ugeskr Laeger. 1998 Nov 23;160(48):6958-61. Danish. PMID 9846090
- [Background] Rowbotham MC. What is a "clinically meaningful" reduction in pain? Pain. 2001 Nov;94(2):131-132. doi: 10.1016/S0304-3959(01)00371-2. No abstract available. PMID 11690725
- [Background] Todd KH, Funk KG, Funk JP, Bonacci R. Clinical significance of reported changes in pain severity. Ann Emerg Med. 1996 Apr;27(4):485-9. doi: 10.1016/s0196-0644(96)70238-x. PMID 8604867
- [Background] Allen RH, Bartz D, Grimes DA, Hubacher D, O'Brien P. Interventions for pain with intrauterine device insertion. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD007373. doi: 10.1002/14651858.CD007373.pub2. PMID 19588429
- [Background] Saav I, Aronsson A, Marions L, Stephansson O, Gemzell-Danielsson K. Cervical priming with sublingual misoprostol prior to insertion of an intrauterine device in nulliparous women: a randomized controlled trial. Hum Reprod. 2007 Oct;22(10):2647-52. doi: 10.1093/humrep/dem244. Epub 2007 Jul 25. PMID 17652452
- [Derived] Akers AY, Harding J, Perriera LK, Schreiber C, Garcia-Espana JF, Sonalkar S. Satisfaction With the Intrauterine Device Insertion Procedure Among Adolescent and Young Adult Women. Obstet Gynecol. 2018 Jun;131(6):1130-1136. doi: 10.1097/AOG.0000000000002596. PMID 29742656
- [Derived] Akers AY, Steinway C, Sonalkar S, Perriera LK, Schreiber C, Harding J, Garcia-Espana JF. Reducing Pain During Intrauterine Device Insertion: A Randomized Controlled Trial in Adolescents and Young Women. Obstet Gynecol. 2017 Oct;130(4):795-802. doi: 10.1097/AOG.0000000000002242. PMID 28885425